CLINICAL TRIAL: NCT01122901
Title: A Phase II and Pharmacodynamic Trial of RO4929097 for Patients With Recurrent/Progressive Glioblastoma
Brief Title: Gamma-Secretase/Notch Signalling Pathway Inhibitor RO4929097 in Treating Patients With Recurrent or Progressive Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped prematurely by Company due to decision to terminate all CTEP supplied drug for further development of RO4929097.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02931; NCI-2012-02931 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000672628; ABTC-0906 (Other: Adult Brain Tumor Consortium); ABTC-0906 (Other: CTEP); U01CA137443 (NIH)
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (gamma-secretase inhibitor RO4929097) (Experimental): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days 1-3, 8-10, 15-17, and 22-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: pharmacological study
- Group B (gamma-secretase inhibitor RO4929097, surgery) (Experimental): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days -6 to -1. Patients undergo surgical resection on day 0. Within 30 days after surgical resection, patients receive gamma-secretase inhibitor RO4929097 as in group A.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given PO
  Other Names: R4733; RO4929097
Procedure: therapeutic conventional surgery — Undergo surgery
  Arms: Group B (gamma-secretase inhibitor RO4929097, surgery)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies
  Arms: Group B (gamma-secretase inhibitor RO4929097, surgery)

SUMMARY:
This phase II trial is studying how well gamma-secretase/Notch signalling pathway inhibitor RO4929097 works in treating patients with recurrent or progressive glioblastoma. Gamma-secretase/Notch signalling pathway inhibitor RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. 6-month progression-free survival (PFS6). (Group A) II. Efficiency of neurosphere generation after pretreatment with RO4929097 (gamma-secretase/Notch signalling pathway inhibitor RO4929097). (Group B)

SECONDARY OBJECTIVES:

I. Radiographic response rate. (Group A) II. Toxicities associated with this regimen. (Group A) III. Overall survival. (Group A) IV. Expression levels of Notch pathway components and downstream targets. (Group B) V. Tumor propagation. An extension of lifespan by 50% in tumor bearing mice (mice bearing fresh tumor tissue). (Group B) VI. Patient event-free survival in correlation with expression levels of Notch pathway components and downstream targets.

VII. 6-month progression-free survival (PFS6). VIII. Toxicities associated with this regimen. IX. Overall survival.

OUTLINE: Patients are assigned to 1 of 2 treatment groups.

GROUP A: Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 orally (PO) once daily (QD) on days 1-3, 8-10, 15-17, and 22-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP B (surgical resection indicated): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days -6 to -1. Patients undergo surgical resection on day 0. Within 30 days after surgical resection, patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 as in Group A.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven glioblastoma which is progressive or recurrent following radiation therapy +/- chemotherapy
* Patients must have measurable contrast-enhancing progressive or recurrent glioblastoma by magnetic resonance imaging (MRI) imaging within two weeks of starting treatment; patient must be able to tolerate MRIs
* GROUP B PATIENTS ONLY: Patients must be eligible for surgical resection according to the following criteria:

  * Expectation that the surgeon can resect >= 50% of the Gd-enhancing tumor with low risk of inducing neurological injury
  * Absence of hematologic, cardiac or other medical contraindications to surgery
  * Surgery must take place Monday-Thursday with the exception of patients being treated at Cleveland Clinic/University Hospitals: these patients may undergo surgery Monday-Friday
  * Patients must have a tumor size >= 2.5 cm in diameter in two perpendicular planes in order to enable correlative studies
  * Paraffin embedded tissue must be available from initial surgical resection at diagnosis (prior to any treatment)
* Patients may have an unlimited number of prior therapy regimens but no prior gamma-secretase inhibitors
* Patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:

  * 3 months from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., small molecule targeted therapy, thalidomide, bevacizumab, etc.)
* Patients may not be on an enzyme-inducing anti-epileptic drug (EIAED); if previously on an EIAED, patient must be off for at least 14 days prior to the first dose of RO4929097
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 4.0 x institutional upper limit of normal
* Creatinine within institutional upper limit of normal OR
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Electrolytes - calcium, chloride, magnesium, potassium, phosphorus, sodium within institutional normal limits
* Patients must be able to provide written informed consent
* Women of childbearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) starting prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately

  * PREGNANCY TESTING: Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days prior to treatment start and be required to agree to have the test repeated within 24 hours prior to the first dose of RO4929097 (serum or urine); a pregnancy test (serum or urine) will also be administered every 4 weeks (within 24 hours prior to starting every cycle) if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing RO4929097, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the potential of RO4929097 to cause serious or life-threatening birth defects
  * Female patients of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had tubal ligation
  * Female patients may be considered to NOT be of childbearing potential for the following reasons:

    * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
    * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
* Patients may not be breast-feeding
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= five years
* Patients must have a Mini Mental State Exam score of >= 15

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety, are ineligible
* Patients with prior treatment with gamma-secretase inhibitors are ineligible
* Patients may not be receiving any other investigational agents
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097 or other agents used in the study are ineligible
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption are ineligible; patients must be able to swallow capsules
* Patients with the following cardiovascular abnormalities are ineligible: baseline QTcF > 450 msec (male) or QTcF > 470 msec (female)
* Patients with a requirement for antiarrhythmics or other medications known to prolong QTc are ineligible
* Patients with a history of being serologically positive for hepatitis B or C, or who have a history of cirrhosis are ineligible
* Patients with a history of uncontrolled hypocalcemia, hypomagnesemia, hyponatremia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, a history of torsades de pointes or other significant cardiac arrhythmias other than chronic stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women or those who are breastfeeding are ineligible
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients who have not recovered to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicities related to prior therapy are not eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, Principal Investigator — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled between April 2011 and May 2012 Patients enrolled in outpatient setting
Groups:
- Group A RO4929097 PO: Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days 1-3, 8-10, 15-17, and 22-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given PO
  pharmacological study: Correlative studies
- Group B RO4929097 Pre Surgery: Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days -6 to -1. Patients undergo surgical resection on day 0. Within 30 days after surgical resection, patients receive gamma-secretase inhibitor RO4929097 as in group A.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given PO
  therapeutic conventional surgery: Undergo surgery
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Group A RO4929097 PO | Group B RO4929097 Pre Surgery
Started | 40 | 7
Completed | 40 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A RO4929097 PO | Group B RO4929097 Pre Surgery | Total
Number analyzed (Participants) | 40 | 7 | 47
Age, Continuous [Median (Full Range); unit: years] | 58 [35 to 75] | 56 [43 to 77] | 57 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 2 | 15
  Male | 27 | 5 | 32
Karnofsky Performance Status Scale [Median (Full Range); unit: units on a scale] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale | 80 [60 to 100] | 80 [60 to 100] | 80 [60 to 100]
Debulking [Count of Participants; unit: Participants] — surgical procedure to remove brain tumor
  Participants
    Yes | 30 | 6 | 36
    No | 10 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Median Progression-free Survival (6-month PFS)
Description: Time to event endpoints for Group A will be measured from the date of first dose. All patients who receive at least one dose of study drug will be included in the analysis. Time to event endpoints for Group B will be measured from the first post-surgical date (this will be considered start date of treatment). Progression defined as: >25% increase sum of products of perpendicular diameters (bi-dimensional measurements) of enhancing lesions (over baseline (BL) if no decrease) on stable or increasing doses of corticosteroids. and/or b) Significant increase in T2/FLAIR nonenhancing lesion on stable or increasing doses of corticosteroids compared to BL scan or best response following initiation of therapy c) Any new lesion. d) Clear clinical deterioration not attributable to other causes apart from the tumor e) Failure to return for evaluation due to death or deteriorating condition.
Time Frame: At 6 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Group A (Post Surgery) & Group B (Pre-surgery) RO4929097 PO: GROUP A Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days 1-3, 8-10, 15-17, and 22-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given PO
  pharmacological study: Correlative studies
  GROUP B Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days -6 to -1. Patients undergo surgical resection on day 0. Within 30 days after surgical resection, patients receive gamma-secretase inhibitor RO4929097 as in group A.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given PO
  therapeutic conventional surgery: Undergo surgery
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Group A (Post Surgery) & Group B (Pre-surgery) RO4929097 PO | Group B RO4929097 Pre Surgery
Number analyzed (Participants) | 40 | 7
months | 1.7 [1.1 to 1.8] | 1.6 [0.8 to 2.3]

2. Primary Outcome: Efficiency of Neurosphere Generation After Pretreatment With RO4929097 (Group B)
Description: This outcome could not be analyzed as the n was too small. The study was terminated prematurely by Hoffman-La Roche Company due to their decision to terminate drug supply for further development of this drug. All CTEP-sponsored trials using RO4929097 were closed to accrual and all patients had to be off treatment by 7/31/12.
Time Frame: At time of surgery
Population: This outcome could not be analyzed as the n was too small. Only had 7 samples. The study was terminated prematurely by Hoffman-La Roche Company due to their decision to terminate drug supply for further development of this drug
Arm/Group | Group B (Gamma-secretase Inhibitor RO4929097, Surgery)
Number analyzed (Participants) | 0

3. Secondary Outcome: Radiographic Response Rate According to the Radiographic Assessment in Neuro-Oncology Criteria (Group A) and Group (B)
Description: RANO:
  Measurable: Bidimensionally measurable lesions w/ clearly defined margins by MRI Evaluable: Unidimensionally measurable lesions, masses w/margins not clearly defined.
  Complete Response (CR): Complete disappearance of all measurable/evaluable disease. No new lesions. No evidence of non-evaluable disease. Patients on minimal/no steroids.
  Partial Response (PR): >/= to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. Responders must be on same/decreasing doses of dexamethasone.
  Stable/No Response: Does not qualify for CR, PR, or progression.
  Progression: 25% increase in the sum of products of all measurable lesions over smallest sum observed (over BL if no decrease), OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Up to 6 months after completion of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A RO4929097 PO | Group B RO4929097 Pre Surgery
Number analyzed (Participants) | 40 | 7
Participants
  Complete Response | 1 | 0
  Partial Response | 0 | 0
  Stable Disease | 3 | 0
  Progression | 33 | 5
  Not Evaluable | 3 | 2

4. Secondary Outcome: Number of Participants With Toxicities Associated With Study Drug (Group A and Group B)
Description: assessed by the National Cancer Institute CTCAE version 4.0 assessed if patient received at least one dose of study drug Grade 3-5 toxicities grade 3 -severe grade 4 - life threatening grade 5 - death
Time Frame: Up to 30 days after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A RO4929097 PO | Group B RO4929097 Pre Surgery
Number analyzed (Participants) | 40 | 7
Participants
  Cognitive Disturbance gr 3 | 1 | 0
  Fatigue gr 3 | 1 | 0
  Hypophosphatemia gr 3 | 4 | 0
  Skin Infection gr 3 | 1 | 0
  AST increase gr 3 | 1 | 0

5. Secondary Outcome: Overall Survival
Description: time to event endpoints for Group A will be measured from date of first dose. All patients who receive at least one dose will be included in analysis.
  Time to event endpoints for Group B will be measured from the first post-surgical date (this will be considered start date of treatment).
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Group A (Post Surgery) RO4929097 PO: GROUP A Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days 1-3, 8-10, 15-17, and 22-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given PO
  pharmacological study: Correlative studies
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given PO
  therapeutic conventional surgery: Undergo surgery
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Group A (Post Surgery) RO4929097 PO | Group B RO4929097 Pre Surgery
Number analyzed (Participants) | 40 | 7
months | 6.6 [5.3 to 10.5] | 6.7 [5.1 to 12]

6. Secondary Outcome: Expression Levels of Notch Pathway Components and Downstream (Group B)
Description: as for outcome 2
Time Frame: At the time of surgery
Population: This outcome could not be analyzed as the n was too small. The study was terminated prematurely by Hoffman-La Roche Company due to their decision to terminate drug supply for further development of this drug.
Arm/Group | Group B (Gamma-secretase Inhibitor RO4929097, Surgery)
Number analyzed (Participants) | 0

7. Secondary Outcome: Tumor Propagation (Group B)
Description: as for outcome 2
Time Frame: At the time of surgery
Population: as for outcome 6
Arm/Group | Group B (Gamma-secretase Inhibitor RO4929097, Surgery)
Number analyzed (Participants) | 0

8. Secondary Outcome: Progression Free Survival
Description: as for outcome 1
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A (Post Surgery) & Group B (Pre-surgery) RO4929097 PO | Group A RO4929097 PO | Group B RO4929097 Pre Surgery
Number analyzed (Participants) | 47 | 40 | 7
months | 1.7 [1.2 to 1.8] | 1.7 [1.1 to 1.8] | 1.6 [0.8 to 2.3]

ADVERSE EVENTS:
Time Frame: 2 year
Arm/Group | Group A RO4929097 PO | Group B RO4929097 Pre Surgery
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/7
Other Adverse Events (participants affected / at risk) | 27/40 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A RO4929097 PO (N=40) | Group B RO4929097 Pre Surgery (N=7)
Alanine aminotransferase increase (Investigations) | 3 (3) | 0 (0)
anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Aspartate aminotransferase increase (Investigations) | 3 (3) | 0 (0)
constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
edema face (General disorders) | 3 (3) | 0 (0)
fatigue (General disorders) | 11 (11) | 1 (1)
electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
platelet count decrease (Investigations) | 4 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
weight loss (Investigations) | 2 (2) | 0 (0)
white blood cell decrease (Investigations) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated prematurely by Company due to their decision to terminate drug supply for further development of this drug. All CTEP-sponsored trials using RO4929097 were closed to accrual and all patients had to be off treatment by 7/31/12.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less